CLINICAL TRIAL: NCT01457027
Title: A Phase IV, Open Label Study to Evaluate the Short and Long Term Immune Response and CROSS-protection After Vaccination With viroSOME Adjuvanted Inflexal V in Elderly Subjects
Brief Title: A Study to Assess Immunogenicity Parameters After Vaccination Against Influenza and to Evaluate How These Parameters Change During the Influenza Season
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INF-V-A007
Record Dates: First submitted 2011-10-20; First posted 2011-10-21 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Immunisation
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Inflexal V

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental)
  Interventions: Biological: Inflexal V

INTERVENTIONS:
Biological: Inflexal V — Inflexal V influenza vaccine, formulated for the WHO requirements ofr the 2011-2012 season, containing per 0.5 mL dose:
  * 15 µg hemagglutinin (HA) antigen of A/California/7/2009 (H1N1)-like virus
  * 15 µg HA antigen of A/Perth/16/2009 (H3N2)-like virus
  * 15 µg HA antigen of B/Brisbane/60/2008-like virus
  Dose: intramuscular administration (M. deltoideus) of a single dose of 0.5 mL on Day 1

SUMMARY:
A study to evaluate the humoral immune response 3 weeks after vaccination with Inflexal V according to the CHMP criteria in elderly subjects for the 2011/2012 WHO recommended vaccine strains, to evaluate immunogenicity parameters 6 months after vaccination for the 3 vaccine strains and to assess the cross-protection against 4 selected circulating heterogeneous A/H1N1 influenza strains 3 weeks after influenza vaccination versus baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adults aged >60 years on the day of enrollment
* Written informed consent
* Females with confirmed menopause (postmenopausal is defined as 12 months with no menses without an alternative medical cause)

Exclusion Criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (≥38.0 °C)
* Prior vaccination with an influenza vaccine for season 2011/2012
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, including oral corticosteroids in dosages of ≥0.5 mg/kg/day prednisolone or equivalent (inhaled or topical steroids are allowed)
* Known immunodeficiency (including leukemia, HIV seropositivity) or cancer
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Participation in another clinical trial
* Employee at the investigational site or relative of the investigator
* Anticipated non-compliance with study procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Seroprotection | 3 weeks after vaccination (Day 22 ± 2 days)
  Seroprotection rate, defined as proportion of subjects with HI antibody titer ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters will be analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Seroconversion | 3 weeks after vaccination (Day 22 ± 2 days)
  Seroconversion rate, defined as proportion of subjects with ≥4-fold increase in HI antibody titer and with a titer of ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters will be analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Geometric Mean Titer | 3 weeks after vaccination (Day 22 ± 2 days)
  GMT of HI antibodies and fold-increase in GMT (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters will be analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)

SECONDARY OUTCOMES:
Geometric Mean Titer | 6 months post-vaccination
  GMT of HI antibodies and fold-increase in GMT (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters will be analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Seroprotection | 6 months post-vaccination
  Seroprotection rate, defined as proportion of subjects with HI antibody titer ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters will be analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Seroconversion | 6 months post-vaccination
  Seroconversion rate, defined as proportion of subjects with ≥4-fold increase in HI antibody titer and with a titer of ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters will be analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Icardi, MD, Principal Investigator — San Martino University Hospital
Locations (1):
- Dept. of Health Sciences, University of Genoa and Hygiene Unit, "San Martino" University Hospital, Genoa, Italy